CLINICAL TRIAL: NCT01734655
Title: Qualitative Evaluation of the Mindful Eating Questionnaire (MEQ) in Pregnant Women
Brief Title: Study of the Validity of Using the MEQ to Measure Mindful Eating in Pregnant Women
Acronym: MEQ
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Corby K. Martin, Associate Professor, Director Ingestive Behavior Laboratory, Pennington Biomedical Research Center
Other Study IDs: PBRC 12013; U01DK094418 (NIH)
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All Participants: Participants will be asked to complete the MEQ, the Eating Inventory Questionnaire, The Mindful Attention Awareness Scale (MAAS), and the Neighborhood Environment Walkability Scale (NEWS). Participants will then be asked to sequentially respond to each of the 28 items and the response choices from the MEQ and briefly discuss their reaction to the items and response choices. Finally, participants will either participate in a focus group or an individual cognitive interview, giving them the opportunity to elaborate on their responses to the MEQ. The first 11 participants completed focus groups and the remaining 29 participants completed individual cognitive interviews.

SUMMARY:
The Specific Aim of this supplemental project is to evaluate the Mindful Eating Questionnaire (MEQ) to determine if it is a valid instrument for pregnant women. During this project, the MEQ will be qualitatively evaluated in a sample of pregnant women who are similar in age, ethnicity, education, and marital status to the women targeted for recruitment in the parent study. The qualitative evaluation will include a focus group with 10 participants followed by 30 individual cognitive interviews. Comments from the interviews will be summarized and analyzed systematically for each of the 28 questions of the MEQ and the interviewer will use findings from initial interviews to inform subsequent interviews. Content validity will be evaluated based on responses from the focus group and cognitive interviews, and MEQ items will be evaluated for comprehension, retrieval, judgment, and response. Strengths, weaknesses, relevance, comprehensiveness, and interpretations will be reported for each of the MEQ questions. We will also have some of the more traditional validation parameters (the inclusion of other questionnaires) in the study to collect data on convergent and discriminant validity. The resulting publication will provide readers with a thorough report on the utility and appropriateness of using the MEQ to quantify mindful eating in pregnant women.

DETAILED DESCRIPTION:
Pre-pregnancy maternal overweight/obesity and excess weight gain during pregnancy are associated with metabolic abnormalities in mothers and their offspring. Despite guidelines developed by the Institute of Medicine (IOM) for appropriate levels of gestational weight gain, more than 50% of overweight and obese pregnant women exceed the recommended amount of weight gain during pregnancy (CDC 2009). Updated guidelines from the Institute of Medicine (IOM) in 2009 suggest that individualized dietary counseling and regular physical activity are necessary for pregnant women to achieve appropriate levels of gestational weight gain (IOM and NRC 2009), yet few studies have examined weight management in overweight pregnant women and none were successful at increasing adherence to the IOM guidelines (Polley, Wing et al. 2002; Olson, Strawderman et al. 2004; Asbee, Jenkins et al. 2009; Shirazian, Monteith et al. 2010; Phelan, Phipps et al. 2011).

This project is a supplement to a parent study called Expecting Success: Personalized management of body weight during pregnancy (U01 DK094418-01 PIs: Leanne M. Redman, Ph.D. & Corby K. Martin, Ph.D.). The parent study will test the efficacy of two interventions at promoting appropriate levels of weight gain during pregnancy compared to each other and to a usual care control group. Appropriate levels of weight gain during pregnancy will be defined by the 2009 IOM gestational weight gain guidelines (CDC 2009). The two interventions include training on mindfulness surrounding eating, hunger, and satiety; hence, it is logical to test if changes in mindfulness differ between the two intervention groups and the usual care group. Moreover, it is possible that change in mindfulness will be associated with the study's outcome or different levels of gestational weight gain between the usual care group and the two intervention groups. Finally, changes in mindfulness could mediate the effect of the two interventions on gestational weight gain.

Despite the possible importance of mindfulness to the eating behavior and weight management of pregnant women, no measure has been validated to measure mindfulness in pregnant women. The Mindful Eating Questionnaire (MEQ) is a 28-item self-report instrument that measures five domains of mindful eating: disinhibition, awareness, external cues, emotional response, and distraction. Mindful eating refers to an unbiased awareness of sensations surrounding eating and although a preliminary study found the MEQ to be a valid measure of mindful eating in healthy adults, it has not been validated in pregnant women. A valid measure of mindful eating is required when an intervention is used to increase mindful eating in pregnant women and evaluate if the increase results in healthier eating habits and effective weight management. Indeed, effectively measuring mindful eating is central to evaluating: 1) if an intervention had the anticipated effect on mindful eating, 2) if increasing mindful eating resulted in changes to eating habits and body mass, and 3) if changes in mindful eating mediated treatment effects.

Relationship of the supplement to the parent grant: Mindfulness training is effective at helping people manage their eating habits, making mindfulness training a viable strategy to use with special populations who struggle with eating and weight management, including pregnant women. During the parent study, two personal weight-management interventions designed to meet the unique needs of pregnant women will be deployed and mindful eating techniques are part of these interventions. Although a preliminary study found the Mindful Eating Questionnaire (MEQ) to be valid in a convenience sample of generally healthy adults, it is not known if the MEQ is an appropriate and valid instrument for use with pregnant women, and the proposed project will answer this question. If the MEQ is valid for use with pregnant women, it can be used in the parent study, as well as other studies, to determine if the interventions are effectively at training participant to mindfully eat and if changes in mindful eating mediate intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age, inclusive
* Overweight or obese at time of conception based on self-report (BMI ≥25 and <40 kg/m2)
* Willingness to participate in either the focus group or the individual interview
* Establish prenatal care by 12 weeks of gestation
* Fluent in the English language; AND
* Singleton pregnancy

Exclusion Criteria:

* Current multiple gestation
* Type I diabetes
* Self-reported gestational diabetes mellitus
* History or current psychotic disorder
* Current major depressive episode, bipolar disorder, or eating disorder
* HIV
* Current smoking, alcohol or drug use
* History of ≥ 3 miscarriages
* Current enrollment in Expecting Success (IRB#11024)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Forty pregnant women (11 will participate in the focus group and 29 will complete individual cognitive interviews) will be recruited who are similar in age, ethnicity, education, and marital status to the women who will be recruited for the parent study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Apolzan JW, Myers CA, Cowley AD, Brady H, Hsia DS, Stewart TM, Redman LM, Martin CK. Examination of the reliability and validity of the Mindful Eating Questionnaire in pregnant women. Appetite. 2016 May 1;100:142-51. doi: 10.1016/j.appet.2016.02.025. Epub 2016 Feb 12. PMID 26879222
- See also: PBRC Web Screener for MEQ — http://www.pbrc.edu/clinical-trials/?studyid=156

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Participants will be asked to complete the MEQ, the Eating Inventory Questionnaire, The Mindful Attention Awareness Scale (MAAS), and the Neighborhood Environment Walkability Scale (NEWS). Participants will then be asked to sequentially respond to each of the 28 items and the response choices from the MEQ and briefly discuss their reaction to the items and response choices in either a focus group format (the first 11 participants) or cognitive interview format (the last 29 participants).
Period: Overall Study
Arm/Group | Participants
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were pregnant women between the ages of 18-40 with a self-reported pre-pregnancy BMI between 25 and 40. All women had a singleton pregnancy and were otherwise healthy.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 40
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m2] | 30.0 (4.1)
Pre-pregnancy Body Weight [Mean (Standard Deviation); unit: kg] | 83.5 (17.6)
Gestational Age [Mean (Standard Deviation); unit: weeks] | 19.9 (8.3)
Current BMI [Mean (Standard Deviation); unit: kg/m2] | 31.8 (4.7)
Current Body Weight [Mean (Standard Deviation); unit: kg] | 86.5 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Test-Retest Reliability of the Mindful Eating Questionnaire (MEQ)
Description: Participants were given the Mindful Eating Questionnaire (MEQ) at their screening visit and study visit in an effort to establish test-retest reliability.
Time Frame: SV and V1; minimum of 24 hours between visits, maximum of 5 months between visits
Measure: Number; unit: test-retest coefficent
Arm/Group | All Participants
Number analyzed (Participants) | 40
test-retest coefficent | .85

2. Primary Outcome: To Determine the Internal Validity of Each of the MEQ's Subscales, we Calculated Cronbach's a
Description: Cronbach's alpha is a measure of internal consistency, that is, how closely related a set of items are as a group. It is considered to be a measure of scale reliability. Alpha coefficients generally range from 0 to 1, with a higher score indicating greater reliability of a scale. However, a "high" value for alpha does not imply that the measure is unidimensional. Technically speaking, Cronbach's alpha is not a statistical test - it is a coefficient of reliability (or consistency).
Time Frame: V1
Population: Pregnant women who were overweight or obese and 18-40 yrs of age.
Measure: Number; unit: Ratio of Variance
Groups:
- All Participants: All Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Ratio of Variance
  Disinhibition | .63
  Awareness | .59
  External Cues | .31
  Emotional Response | .59
  Distraction | .68

3. Primary Outcome: Convergent Validity of the Mindful Eating Questionnaire Compared to the Eating Inventory (EI) Restraint Subscale
Description: The convergent validity of the Mindful Eating Questionnaire was assessed using the Eating Inventory (EI) subscales (restraint, disinhibition, hunger) by calculating Pearson correlation coefficients. Below are the results for the comparison of the Mindful Eating Questionnaire's subscales to the Eating Inventory restraint subscale. Correlations were run with and without the External Cues subscale (ECS) since it was found not to be internally consistent.
Time Frame: V1
Population: Pregnant women who were overweight or obese and 18-40 yrs of age.
Measure: Number; unit: correlation coefficients
Arm/Group | All Participants
Number analyzed (Participants) | 40
correlation coefficients
  Disinhibition** | .46
  Awareness | .07
  External Cues | -.07
  Emotional Response** | .48
  Distraction | .26
  Total Score (w ECS) | .40
  Total Score (w/o ECS)** | .46
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p < .01, correlation analysis

4. Primary Outcome: Convergent Validity of the Mindful Eating Questionnaire Subscales to the Eating Inventory Disinhibition Subscale
Description: The convergent validity of the Mindful Eating Questionnaire was assessed using the Eating Inventory subscales by calculating the Pearson correlation coefficients. Below are the results for the comparison of the Mindful Eating Questionnaire's subscales to the Eating Inventory Subscale of Disinhibition. Correlations were run with and without the External Cues subscale since it was found not to be internally consistent.
Time Frame: V1
Measure: Number; unit: correlation coefficients
Groups:
- Participants: Participants will be asked to complete the MEQ, the Eating Inventory Questionnaire, The Mindful Attention Awareness Scale (MAAS), and the Neighborhood Environment Walkability Scale (NEWS). Participants will then be asked to sequentially respond to each of the 28 items and the response choices from the MEQ and briefly discuss their reaction to the items and response choices. Finally, participants will either participate in a focus group or an individual cognitive interview, giving them the opportunity to elaborate on their responses to the MEQ. The first 11 participants completed focus groups and the remaining 29 participants completed individual cognitive interviews.
Arm/Group | Participants
Number analyzed (Participants) | 40
correlation coefficients
  Disinhibition** | -.64
  Awareness | -.30
  External Cues | -.04
  Emotional Response** | -.68
  Distraction | -.33
  Total Score (w ECS)** | -.65
  Total Score (w/o ECS)** | -.70
Statistical Analysis 1: Comparison: Participants; Test type: Superiority or Other; p < .01, correlation analysis

5. Primary Outcome: Convergent Validity of the MEQ Subscales Compared to the EI Hunger Subscale
Description: The convergent validity of the Mindful Eating Questionnaire was assessed using the Eating Inventory subscales of restraint, disinhibition and hunger by calculating the Pearson correlation coefficients. Below are the results for the comparison of the Mindful Eating Questionnaire's subscales to the Eating Inventory Subscale of Hunger. Correlations were run with and without the External Cues subscale since it was found not to be internally consistent.
Time Frame: V1
Measure: Number; unit: correlation coefficients
Arm/Group | Participants
Number analyzed (Participants) | 40
correlation coefficients
  Disinhibition** | -.54
  Awareness | -.04
  External Cues | -.01
  Emotional Response** | -.41
  Distraction | -.40
  Total Score (w ECS)** | -.46
  Total Score (w/o ECS)** | -.51
Statistical Analysis 1: Comparison: Participants; Test type: Superiority or Other; p < .01, correlation analysis

6. Primary Outcome: Correlation of the MEQ Subscales to the MAAS
Description: The convergent validity of the MEQ was also assessed by calculating the pearson correlation between the MEQ subscales and the Mindful Attention Awareness Scale (MAAS). Correlations were run with and without the External Cues subscale since it was found not to be internally consistent. **Indicates correlation significant at the .01 level
Time Frame: V1
Measure: Number; unit: correlation coefficients
Arm/Group | Participants
Number analyzed (Participants) | 40
correlation coefficients
  Disinhibition** | .40
  Awareness | .245
  External Cues | .01
  Emotional Response** | .44
  Distraction** | .64
  Total Score (w ECS)** | .58
  Total Score (w/o ECS)** | .63

ADVERSE EVENTS:
Groups:
- All Participants: Pregnant women who were overweight or obese and 18-40 yrs of age.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=40)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — A participant reported that she had experienced some abdominal pain. This was determined to be non-serious and unrelated to the study by the medical investigator.
Vaginal Spotting (Pregnancy, puerperium and perinatal conditions) | 1 (1) — A participant reported that she had experienced some vaginal spotting. She visited her OB/GYN and it was determined to be harmless. This was determined to be non-serious and unrelated to the study by the medical investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No